CLINICAL TRIAL: NCT04541082
Title: A First-in-human Phase I Single-agent Dose-escalation, Food Effect and Dose Expansion Study of Oral ONC206 in Recurrent and Rare Primary Central Nervous System Neoplasms
Brief Title: Phase I Study of Oral ONC206 in Recurrent and Rare Primary Central Nervous System Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC206-001; NIH 20C0069 (Other: National Institutes of Health)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma, Adult; Anaplastic Oligodendroglioma; Anaplastic Astrocytoma; Pilocytic Astrocytoma; Oligodendroglioma; Gliomatosis Cerebri; Pleomorphic Xanthoastrocytoma; Anaplastic Pleomorphic Xanthoastrocytoma; Diffuse Midline Glioma, H3 K27M-Mutant; Ependymoma; Ependymoma, Anaplastic; Medulloblastoma; Teratoid Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Neuroectodermal Tumors; Anaplastic Meningioma; Atypical Meningioma; Choroid Plexus Neoplasms; Pineal Tumor; Diffuse Astrocytoma; Glial Tumor
Keywords: Glioblastoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Diffuse Astrocytoma; Oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Oligodendroglioma; Astrocytoma; Neoplasms, Neuroepithelial; Ependymoma; Medulloblastoma; Typical Teratoid Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Neuroectodermal Tumors; Meningioma; Choroid Plexus Neoplasms; Pinealoma; Glioma | interventions — ONC206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ONC206 (Experimental)
  Interventions: Drug: ONC206

INTERVENTIONS:
Drug: ONC206 — ONC206 is a member of the imipridone class of anti-cancer small molecules that share a unique tri-heterocyclic core chemical structure and target G protein-coupled receptors.

SUMMARY:
The primary objective of this Phase 1, open-label, dose-escalation, and exploratory study is to evaluate the safety and tolerability profile (establish the maximum-tolerated dose) and evaluate the occurrence of dose-limiting toxicities (DLTs) following single weekly or multiple-day weekly dose regimens of single-agent, oral ONC206 in patients with recurrent, primary central nervous system (CNS) neoplasms.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation, and exploratory study of ONC206 in patients with recurrent, primary CNS neoplasms. All patients will be informed about the study and potential risks and required to provide written informed consent prior to undergoing study-related procedures.

There will be a total of 11 Dose Levels. Dose-escalation for Dose Levels 1 through 5 proceeded according to standard 3+3 design using a 28-day DLT window. The first cohort of 3 patients enrolled into the study received Dose Level 1 followed by increments as per the modified Fibonacci sequence. It is anticipated that approximately 46 patients will be enrolled in order to determine the MTD of ONC206.

For Dose Levels 1 through 5, a safety evaluation was conducted when 3 evaluable patients have completed 1 cycle (28 days) of therapy. After Protocol Amendment 6, all available PK data will also be considered for dose escalation decisions. Dose levels may be adjusted based on review of PK data but will not exceed maximum dose levels described in Table 6. Additionally, dose frequencies (e.g., once daily or 3 times daily) may be added and/or removed based on emerging PK data and concentration projections.

Prior to advancing/changing dose levels, a cohort summary must be completed and submitted to the sponsor Medical Monitor, for review and approval. Dose escalation for subsequent patients will proceed as follows:

* If no DLT is reported at a dose level, that dose level will be considered safe, and patient(s) will be enrolled at the next dose level. Toxicity information will continue to be evaluated from the time of the first protocol specific intervention, until 30 days from the last dose of study drug.
* If 1 patient in a cohort of 1 experiences a DLT, the dose level will be expanded to obtain an additional 2 evaluable patients.
* If 1 patient in a cohort at a dose level experiences a DLT, the dose level will be expanded to obtain an additional 3 evaluable patients.
* If 2 of 3 patients in a cohort at a dose level experience a DLT, that dose level will not be considered safe, no further dose escalation will take place, and the MTD will have been exceeded*.
* If 1 patient experiences a DLT among the expanded cohort of evaluable patients, a cohort of 3 patients will be enrolled in the next higher dose level.
* If 2 or more patients experience a DLT among the expanded cohort of evaluable patients, that dose level will not be considered safe, no further dose escalation will take place, and the MTD will have been exceeded*. The previous dose level at which ≤1 patients experienced a DLT will be declared the MTD.

  * When the MTD has been exceeded:

If less than 6 patients have been treated in the next lower dose level (the possible MTD level), additional patients will be entered into this dose level until there are 6 patients treated. If ≤1 of these 6 patients encountered DLT, then this dose level will be declared to be the MTD. If 2 or more of the 6 patients encounter DLT, then the MTD has been exceeded.

Given the experience with ONC201, it is possible a MTD may not be reached through the planned dose escalation cohorts. If the therapeutic target concentrations have been achieved in the dose escalation cohorts, and no DLT has been identified, then analysis of the safety and PK data will be evaluated by the Investigators and the Sponsor. Further dose levels may then be considered at higher intermittent dosing schedules and will be added by protocol amendment with review by the Institutional Review Board (IRB) before implementation.

Toxicities will be graded using the Common Terminology Criteria for Adverse Events Version 24.0 (CTCAE 24.0). If the CTCAE 24.0 does not apply to an adverse event, it will be graded as mild, moderate, or severe.

DLTs will be assessed during the first course of each cohort (28 days), and refers to a study drug related or possibly related event that meets 1 of the following criteria using the NCI CTCAE version 5.0:

* Grade 3 or higher non-hematologic toxicity.
* Grade 4 hematologic toxicity (ANC <0.5 × 109/L and platelet count <25 × 109/L). Lymphopenia is not considered a DLT. A confirmed DLT requires 2 consecutive measurements separated by 48 hours.
* Grade 3 neutropenia (ANC <1.0 × 109/L) with elevated fever (>101°F). A confirmed DLT requires 2 consecutive measurements.
* Grade 3 thrombocytopenia with clinically significant bleeding.
* Inability to receive the scheduled Cycle 2, Day 1 dose of study drug within 14 days due to study drug-related toxicity persisting from Cycle 1 or study drug-related toxicity newly encountered on Day 1 of Cycle 2.

Safety and tolerability will be monitored by assessing physical examinations including height (at Screening only) and weight, KPS, vital signs, ECG, laboratory assessments including hematology, chemistry, and coagulation, as well as collecting of the AEs at every visit.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to participate in the study:

1. Patients aged ≥18 years with a recurrent, primary CNS neoplasm. For all cohorts, patients must have a histologically confirmed primary CNS neoplasm. Primary CNS neoplasms in this study include, but are not limited to, the following: glioblastoma and glioblastoma histologic subtypes, gliosarcoma, primary CNS sarcomas, anaplastic glial neoplasms including anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed neuronal-glial tumors, and pilocytic astrocytoma with anaplastic features, diffuse astrocytoma, oligodendroglioma, gliomatosis cerebri, pleomorphic xanthoastrocytoma, anaplastic pleomorphic xanthoastrocytoma, diffuse midline gliomas and histone mutated gliomas (NOTE: Patients with H3 K27M-mutant diffuse gliomas are excluded unless the primary tumor is located in the pons or spinal cord, or the patient has completed front line radiation or received ONC201 therapy prior to 01 January 2023), ependymoma, anaplastic ependymoma, and all ependymoma subtypes, medulloblastoma and all medulloblastoma subtypes, atypical teratoid/rhabdoid tumor, primary CNS embryonal/primitive neuroectodermal tumors, atypical and anaplastic meningiomas, choroid plexus tumors, and pineal region tumors.
2. Patients must have recurrent and measurable disease as defined by RANO criteria, using either the HGG and/or LGG RANO criteria based on tumor type, after having received established standard of care treatment for their disease and have no standard treatment options available as determined by the investigators. There is no limit on the number of total recurrences or prior therapies. However, prior therapies with known clinical benefit (including radiation) for specific tumor types are required. If patients are deemed ineligible for such therapies in the opinion of the Investigator, the Investigator must document the reason the patient is considered ineligible.
3. Patients must have a Karnofsky Performance Score (KPS) of greater than or equal to 70. Patients with severe paraparesis/paraplegia who need minimal assistance for self-care due to their motor deficit but are otherwise functionally independent will be considered eligible.
4. (Inclusion Criterion #4 was removed in Amendment 3.)
5. Patients must not have received prior investigational or approved cytotoxic chemotherapy within 28 days prior to the first dose of study drug (Cycle 1, Day 1); 42 days in the case of nitrosoureas; 42 days in the case of bevacizumab; 28 days or 5 half-lives (whichever is less; but not less than 14 days) in case of investigational or approved molecularly targeted agent; 14 days in the case of radiotherapy.
6. (Inclusion Criterion #6 was removed in Amendment 7.)
7. Patients with AEs Grade ≥2 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must have all their AEs resolved prior to the first dose of study drug (Cycle 1, Day 1), except for alopecia or neuropathy; Grade 1 or 2 lymphopenia is allowed.
8. Patients must not have undergone major surgery 4 weeks prior to the first dose of study drug (Cycle 1, Day 1) and must have completely recovered from any surgery (minor surgical procedures such as skin biopsies and port placement done on an outpatient basis do not require a waiting period).
9. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) ≥1,500/mcL.
   * Platelets ≥100,000/mcL.
   * Hemoglobin ≥9.0 mg/dL without transfusion in 2 prior weeks.
   * Total bilirubin ≤1.5 × upper limit of normal (ULN) (patients with Gilbert's syndrome may be included with total bilirubin >1.5 × ULN if direct bilirubin is ≤1.5 × ULN).
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5 × ULN.
   * Measured or estimated creatinine clearance (CLcr) ≥40 mL/minute for patients with creatinine levels above normal. CLcr will be calculated by the Cockcroft-Gault equation for renal function.
10. (Inclusion Criterion #10 was removed in Amendment 3)
11. Patients must provide a tumor specimen (paraffin-embedded block and/or frozen tissue) from a prior resection or biopsy available that is sufficient to perform biomarker assays, ≥15 unstained slides for immunohistochemistry (IHC) analysis must be received by the NOB by the first dose of study drug (Cycle 1, Day 1). For patients with ≥10 to <15 slides, eligibility will be reviewed on a case-by-case basis.
12. Dependent upon dose level assignment and drug formulation (i.e., capsules versus powder in bottle [PIB]), patients must be able to either swallow oral capsules or swallow liquids.
13. Patients must provide study-specific informed consent prior to enrollment. No Durable Power of Attorney or Next of Kin can provide initial consent.
14. Patients must be able to tolerate a magnetic resonance imaging (MRI) study with intravenous gadolinium contrast.
15. (Inclusion Criterion #15 was removed in Amendment 6)
16. Patients must have a negative COVID-19 test within 72 hours of the first dose of study drug (Cycle 1, Day 1). Patients who had documented COVID-19 infection within 90 days of treatment but more than 20 days from infection do not need to be tested.
17. (Inclusion Criterion #17 was removed in Amendment 6)

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. (Exclusion Criterion #1 was removed in Amendment 3)
2. Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC206 (e.g., ONC201) or its excipients.
3. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
4. Patients who are unable or unwilling to abide by the study protocol or cooperate fully with the Investigator.
5. Patients with a known HIV-positive test on combination anti-retroviral therapy are ineligible for this initial first-in-human trial because of the potential for PK interactions with ONC206.
6. Patients with active cardiac disease, including any of the following:

   * Corrected QT interval (QTc) ≥470 msec on screening electrocardiogram (ECG; using the QTc by Fridericia's [QTcF] formula);
   * Angina pectoris that requires the use of anti-anginal medication;
   * Ventricular arrhythmias except for benign premature ventricular contractions;
   * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication;
   * Conduction abnormality requiring a pacemaker;
   * Valvular disease with documented compromise in cardiac function; and/or
   * Symptomatic pericarditis.
7. Patients with a history of cardiac dysfunction including any of the following:

   * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular ejection fraction function;
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV); and/or
   * Documented cardiomyopathy.
8. Patients who have had an ischemic or hemorrhagic stroke in the last 3 months. If the patient has had a recent tumor resection, cerebral ischemic or hemorrhagic changes that occur peri operatively are not an exclusion.
9. Patients with refractory epilepsy are excluded. Patients with primarily or secondarily generalized seizures in the 28 days prior to study enrollment will be excluded. Peri-operative seizures, defined as seizures occurring within the 7 days after a stereotactic biopsy, open biopsy, or surgical resection will not be an exclusion as long as the patient has had no generalized seizures starting 8 days after the surgical procedure. Patients with prior seizures must be on stable doses of 1 or 2 seizure medications for at least 14 days prior to study enrollment.
10. Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of ONC206 (uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
11. Patients who have been treated with any hematopoietic colony-stimulating growth factors (CSFs) (e.g., granulocyte-CSF, granulocyte-macrophage-CSF) ≤2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued.
12. Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin derivative anticoagulant.
13. Patients who are taking strong inhibitors or inducers of cytochrome P450 (CYP) 3A4, 2D6, 1A2, 2C9, and 2C19 within at least 14 days prior to the first dose of study drug (Cycle 1, Day 1); these medications are excluded throughout the study.
14. Women who are pregnant or breast feeding.
15. Women of child-bearing potential with a positive serum pregnancy test ≤72 hours prior to the first dose of study drug (Cycle 1, Day 1).
16. Patients who are receiving concomitant standard and/or investigational anti-cancer therapy.
17. Patients with alcohol or substance abuse which, in the opinion of the Investigator, would interfere with compliance or safety.
18. Patients with the presence of any other serious and/or unstable pre-existing medical disorder, psychiatric disorder, or other conditions that could interfere with patients' safety, obtaining informed consent or compliance to the study procedures as determined by the Investigators.
19. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, or men who do not agree to use highly effective contraception during treatment and for 16 additional weeks after the final dose of study drug.

    Highly effective contraception is defined as either:
    * True abstinence: When this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Sterilization: Females must have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female patients on the study, the vasectomized male partner should be the sole partner for that patient.
    * If patients are not practicing true abstinence and/or if the patient or sexual partner have not had a sterilization procedure as listed above, patients and their sexual partners must follow double barrier contraception in accordance with the guidelines for contraception below:

      * Females of childbearing potential:

        * Must use an intrauterine device or intrauterine system, during dosing of any study agent and for 16 weeks after final dose of study drug; or
        * Must use a double barrier method of contraception: use of an occlusive cap (diaphragm or cervical/vault cap) with spermicide for women combined with use of a condom by their male partners capable of conceiving offspring.
      * Males capable of conceiving offspring must use condoms during dosing of study agent and for an additional 16 weeks after final dose of study drug.

    Note: Oral, implantable, or injectable contraceptives may be affected by CYP interactions, and are therefore not considered effective for this study.
20. Previous receipt of ONC201, placebo, or blinded study drug from an ONC201 clinical study, or from any other source for H3 K27M-mutant diffuse glioma on or after 01 January 2023.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of single-agent, oral ONC206 | 28 Days
  MTD was determined by testing increasing doses up to 200 mg twice daily for 3 successive days a week.
  MTD reflects the highest dose of drug that did not cause a Dose-Limiting Toxicity (DLT) in >33% of participants. DLTs will be assessed in the first course of each cohort (28 days), and refer to a study drug-related or possibly related event that meets 1 of the following criteria defined in the subsequent Primary Outcome Measure using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE 5.0).
Number of Participants who Experienced Dose-Limiting Toxicities (DLTs) | 28 Days
  DLTs will be assessed in the first course of each cohort (28 days), and refer to a study drug-related or possibly related event that meets 1 of the following criteria using NCI CTCAE 5.0:
  * Grade 3 or higher non-hematologic toxicity.
  * Grade 4 hematologic toxicity (ANC <0.5 × 109/L and platelet count <25 × 109/L). Lymphopenia is not considered a DLT. A confirmed DLT requires 2 consecutive measurements separated by 48 hours.
  * Grade 3 neutropenia (absolute neutrophil count [ANC] <1.0 × 109/L) with elevated fever (>101°F). A confirmed DLT requires 2 consecutive measurements.
  * Grade 3 thrombocytopenia with clinically significant bleeding.
  * Inability to receive the scheduled Cycle 2, Day 1 dose of study drug within 14 days due to study drug-related toxicity persisting from Cycle 1 or study drug-related toxicity newly encountered on Day 1 of Cycle 2.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Nguyen TTT, Shang E, Schiffgens S, Torrini C, Shu C, Akman HO, Prabhu VV, Allen JE, Westhoff MA, Karpel-Massler G, Siegelin MD. Induction of Synthetic Lethality by Activation of Mitochondrial ClpP and Inhibition of HDAC1/2 in Glioblastoma. Clin Cancer Res. 2022 May 2;28(9):1881-1895. doi: 10.1158/1078-0432.CCR-21-2857. PMID 35417530